CLINICAL TRIAL: NCT02954068
Title: Intravenous Versus Intramuscular Administration of Oxytocin and Its Relationship With Postpartum Bleeding and Other Clinical Signs: a Randomized Placebo-controlled Study
Brief Title: IV Versus IM Administration of Oxytocin for Postpartum Bleeding
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: Centro Rosarino de Estudios Perinatales (CREP) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 3008
Record Dates: First submitted 2016-10-28; First posted 2016-11-03 (Estimated); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Postpartum Hemorrhage
Keywords: Oxytocin
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- IV Infusion (Active Comparator): Oxytocin 10 IU, 500 ml IV infusion within 40 minutes + intra muscular injection of placebo, 10 IU
  Interventions: Drug: IV Oxytocin + IM placebo
- IM administration (Active Comparator): Oxytocin 10 IU via intra muscular injection + Intravenously administered placebo, 10 IU, 500ml
  Interventions: Drug: IM Oxytocin + IV placebo

INTERVENTIONS:
Drug: IV Oxytocin + IM placebo
  Arms: IV Infusion
Drug: IM Oxytocin + IV placebo
  Arms: IM administration

SUMMARY:
This double-blind, randomized controlled trial will evaluate the effect of the route of administration of 10 IU of oxytocin on the average blood loss postpartum. Participants will be randomized to receive 10 IU of oxytocin by IV infusion or 10 IU of oxytocin by injection IM

ELIGIBILITY:
Inclusion Criteria:

* She is present to give birth to a live fetus
* Vaginal delivery
* Willing to participate in the study
* Able to give informed consent

Exclusion Criteria:

* Scheduled for a cesarean
* Reject the placement of an IV during labor (for intravenous infusion)
* Cannot give informed consent for any reason
* Not willing and / or cannot answer questions about background

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 543 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Amount of blood loss (mL) | 1 hour postpartum
Proportion of women who had postpartum blood loss ≥500 ml | 1 hour postpartum

SECONDARY OUTCOMES:
Proportion of women who had postpartum blood loss ≥1000 ml | 1 hour postpartum
Average change in hemoglobin level | pre-delivery and at least 24 hours postpartum
Average time required until expulsion of the placenta | 1 hour postpartum
Proportion who needed additional Interventions | Through study completion, an average of 24-48 hours postpartum
Side effects | 1 hour postpartum
Blood pressure | 15, 30, 45 and 60 minutes postpartum
Heart rate | 15, 30, 45 and 60 minutes postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects; Ilana Dzuba, MPH, Principal Investigator — Gynuity Health Projects; Guillermo Carroli, MD, Principal Investigator — Centro Rosarino de Estudios Perinatales (CREP)
Locations (1):
- Hospital J.R. Vidal, Corrientes, Argentina

REFERENCES:
- [Derived] Oladapo OT, Okusanya BO, Abalos E, Gallos ID, Papadopoulou A. Intravenous versus intramuscular prophylactic oxytocin for the third stage of labour. Cochrane Database Syst Rev. 2020 Nov 9;11(11):CD009332. doi: 10.1002/14651858.CD009332.pub4. PMID 33169839